CLINICAL TRIAL: NCT00925756
Title: The Impact of CCR5 Inhibitor Treatment Intensification on CD4+ T-cell Recovery and Gene Expression Profiles in HIV-Infected Patients With Viral Suppression
Brief Title: CCR5 Inhibitor Treatment Intensification on CD4+ T-cell Recovery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of California, Los Angeles (Other); University of Southern California (Other); Pfizer (Industry); California HIV/AIDS Research Program (Other)
Responsible Party: Principal Investigator, Sheldon Morris, Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTG 590
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: HIV Infections
Keywords: HIV; low CD4 recovery; Low CD4 recovery despite HIV control; Treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Maraviroc 150 mg, 300 mg, or 600 mg twice daily (Experimental): This was a single arm study where Maraviroc was added for 24 weeks.
  Maraviroc was dose-adjusted for concomitantly administered HIV medications according to the manufacture's recommendations:
  150 mg twice daily with strong CYP3A4 inhibitors, including:
  * Protease inhibitors (except tipranavir/ ritonavir)
  * Delavirdine
  * ketoconazole, itraconazole, clarithromycin, nefazadone, telithromycin
  * Darunavir/r + etravirine
    300 mg twice daily with non-inducers/ non-inhibitors of CYP3A4, including:
  * Tipranavir/ ritonavir
  * Nevirapine
  * All NRTIs
  * Enfuvirtide
    600 mg twice daily with strong CYP3A4 inducers, including:
  * Efavirenz, etravirine
  * rifampin
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — Maraviroc will be given dose-adjusted to background HIV treatment (150 mg, 300 mg, or 600 mg twice daily)
  Other Names: Selzentry

SUMMARY:
CCTG 590 is a open-label study to evaluate the impact of therapy intensification with Maraviroc (MVC) (a CCR5 inhibitor) to a stable suppressive HIV antiretroviral regimen on the rate of CD4+ T-cell recovery and gene expression profiles. Patients on a stable first-line HIV regimen with continued viral suppression and sub-optimal CD4+ T-cell counts will be eligible for this study. Those who are found to be eligible will have MVC (dose-adjusted to background HIV regimen) added to their current HIV regimen for 24 weeks. After the 24 week intensification, the MVC will be discontinued, the original antiretroviral regimen will be continued and the subjects will be followed for an additional 12 weeks.

The investigators hypothesize that MVC will improve the rate of CD4 recovery. This improved CD4 recovery will be associated with favorable changes in gene expression profiles of genes involved with CD4 maintenance and circulation.

DETAILED DESCRIPTION:
Blunted CD4+ T-cell responses during viral control may be a consequence of on-going T-cell destruction in the regenerative phase of CD4 recovery from activation-induced apoptosis and/or reduced production from decreased thymic output. Maraviroc, a CCR5 inhibitor, may improve the clinical status of HIV-infected by two distinct mechanisms. First, by blocking HIV entry into CD4+ T-cells, CCR5 inhibitors have direct antiviral activity. Second, as the pro-inflammatory state of HIV infection up-regulates CCR5 ligands and receptors, this CCR5 receptor antagonist may abrogate immune activation and resultant T-cell apoptosis. Importantly, MVC binds CCR5 receptors without inducing intracellular signaling or altering cell-surface expression. Potentially, MVC intensification during viral suppression with ART may further decrease persistent activation-induced apoptosis and improve repair and remodeling of lymphoid tissue leading to increased CD4+ T-cell recovery and function.

The aim of this study is to evaluate a potentially therapeutic immunomodulatory effect of MVC. Several measures of immune homeostasis will be determined in this study, including functional genomic analysis and extended T-cell phenotyping. Genes responsive to MVC therapy will be identified and categorized into functional groups. Based upon existing literature of the identified genes and observed immune responses (change in CD4/CD8 subsets) during MVC therapy, a model of CCR5 responsive-genes and potential impact on immune recovery will be outlined. Potentially, individuals experiencing immune discordance during suppressive ART may be better treated by MVC antiretroviral intensification.

1. We hypothesize that expression will decrease among genes involved in immune activation (NF-kB, MAPK, nuclear factor of activated T-cells, MYD88 and STAT1), apoptosis (Fas ligand and TRAIL) and trafficking/repopulation of T-cells (CCR5, MIP-1α, MIP-1β and RANTES) and increase among genes involved in tissue repair (platelet-derived growth factor, insulin-like growth proteins and osteoblast-specific transcription factor).

1. The gene expression profiles induced by MVC will be associated with a favorable increase in the rate of CD4+ T-cell recovery.
2. The rate of CD4 recovery (cells/month) will be greater during MVC compared to before.
3. The proportion of cells expressing activation/ apoptosis markers will decrease from baseline and this decrease will be associated with improved CD4 recovery.
4. The proportion of naïve cells will increase from baseline and this increase will be associated with improved CD4 recovery.
5. The rate of CD4 recovery will be greater among those subjects receiving PI-containing treatment regimens compared to those receiving NNRTI-containing treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection
2. All available CD4+ T cell counts within the last 12 months of screening below 350 cells/mm3 (minimum of 3 values obtained > 30 days apart).
3. HIV treatment with a stable (for at least 6 months) antiretroviral regimen consisting of at least 2 NRTIs and either a protease inhibitor boosted with low dose ritonavir or an NNRTI. A stable regimen is defined as no additions or deletions for more than 14 cumulative days.
4. Patient considered to be receiving initial HIV regimen (history of medication substitution for toxicity is allowed).
5. All available plasma HIV RNA levels within the last 12 months are below the level of detection. Isolated values that are detectable but < 1000 copies will be allowed as long as the plasma HIV RNA levels before and after this detectable time point are undetectable - The subject should have a minimum of 3 values obtained > 30 days apart.
6. Females of childbearing potential must have a negative serum pregnancy test at screening and agree to use a double-barrier method of contraception throughout the study period.
7. Men and women age ≥ 18 years.

Exclusion Criteria:

1. Current antiretroviral regimen contains tenofovir disoproxil fumarate AND didanosine in combination.
2. History of chronic hepatitis C (defined as HCV antibody positive and HCV RNA detectable).
3. History of chronic active hepatitis B (defined as surface antibody negative, surface antigen positive and HBV DNA detectable).
4. Concurrent use of G-CSF or GM-CSF.
5. Prior or concurrent use of IL-2.
6. Prior or concurrent use of a CCR5 inhibitor.
7. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
8. Use of any immunomodulator, HIV vaccine, or investigational therapy within 30 days of study entry.
9. Use of human growth hormone within 30 days prior to study entry.
10. Initiation of testosterone or anabolic steroids within 30 days prior to study entry. (Exception: Chronic replacement dosages in patient's with diagnosed hypogonadism is allowed).
11. Evidence of splenic sequestration or suppressed bone marrow function:

    * Clinical or radiographic evidence of significant splenomegaly.
    * History of leukemia or lymphoma.
    * History of myelosuppressive chemotherapy or irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-10-20 (Actual); Primary Completion 2012-05-02 (Actual); Study Completion 2014-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Morris, MD, Study Chair — UC San Diego AntiViral Research Center (AVRC); Richard Haubrich, MD, Principal Investigator — University of California, San Diego
Locations (3):
- United States (3):
  - University Southern California, Los Angeles, California
  - University California San Diego, San Diego, California
  - Harbor-UCLA, Torrance, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Maraviroc Intensification: Maraviroc will be added to patient's existing HIV treatment regimen dose-adjusted to background HIV medications
  Maraviroc: Maraviroc will be given dose-adjusted to background HIV treatment
Period: Overall Study
Arm/Group | Maraviroc Intensification
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Maraviroc Intensification
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, not Hispanic | 7
  Black | 2
  White Hispanic | 21
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Differences in Gene Expression Profiles Obtained at Baseline and Week 4 and Week 24.
Description: To determine differential gene expression in T-Cells due to MVC exposure between week 0, 4 and 24 weeks.
  Repeated measures (RM) ANOVA was used to identify genes whose expression changed over the course of MVC administration. Multivariate permutation tests under default settings (80% confident no more than 10% false positives) were performed using BRB-Array Tools. Gene assignment to temporal profiles was performed using a non- parametric clustering algorithm in Short Time-series Expression Miner (STEM)
Time Frame: Baseline to Week 24
Population: 32 participants received intervention and were followed for CD4+ counts. 25 of 32 participants had microarray analysis done.
Measure: Number; unit: -fold TNF downregulation
Arm/Group | Maraviroc Intensification
Number analyzed (Participants) | 25
-fold TNF downregulation | 1.44

2. Secondary Outcome: CD4+ T-cell Absolute Count and Percentage at Baseline, Weeks 4 and 24.
Description: To compare the CD4+/CD8+ T-cell absolute count and percentage change at Weeks 4 and 24 from Baseline. Wilcoxon signed rank test was used to assess changes in T cell counts, percentages, CD4+ T cell recovery slopes and changes in T cell phenotypes measured by flow cytometry.
Time Frame: Baseline to Week 24
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Maraviroc Intensification
Number analyzed (Participants) | 32
cells/mm^3
  Wk 4 CD4+ cells (absolute) | 6.50 [-21.5 to 32.88]
  Wk 4 CD8+ cells (absolute) | 46 [-41.5 to 96.0]
  Wk 24 CD4+ cells (absolute) | 36.75 [16.75 to 64.12]
  Wk 24 CD8+ cells (absolute) | 100.00 [3.25 to 178.88]

3. Secondary Outcome: Change in CD4+/CD8+ T-cell Immune Activation, Maturation, Regulatory and Apoptosis Markers at Baseline and Weeks 4 and 24.
Description: To compare the percent change of CD4+/CD8+ T-cell
Time Frame: Baseline to Week 24
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Maraviroc Intensification
Number analyzed (Participants) | 32
cells/mm^3
  Wk 4 CD4+ total | 0.62 [-0.61 to 1.21]
  Wk 4 CD4+ naive | -0.47 [-1.64 to 0.99]
  Wk 4 CD4+ central memory | 0.43 [-1.56 to 4.98]
  Wk 4 CD4+ effector memory | -0.33 [-1.81 to 1.00]
  Wk 4 CD4+ effector | 0.00 [-0.10 to 0.06]
  Wk 4 CD4+ immune senescence | -0.12 [-1.16 to 0.46]
  Wk 24 CD4+ total | 1.12 [-0.55 to 2.64]
  Wk 24 CD4+ naive | 0.52 [-0.98 to 2.49]
  Wk 24 CD4+ central memory | -0.15 [-2.98 to 2.78]
  Wk 24 CD4+ effector memory | -0.30 [-2.04 to 0.84]
  Wk 24 CD4+ effector | 0.00 [-0.15 to 0.15]
  Wk 24 CD4+ immune senescence | -0.25 [-0.78 to 0.74]
  Wk 4 CD8+ total | 0.90 [-0.92 to 2.84]
  Wk 4 CD8+ naive | -0.45 [-2.32 to 0.59]
  Wk 4 CD8+ central memory | 0.83 [-0.16 to 2.26]
  Wk 4 CD8+ effector memory | 0.73 [-0.64 to 3.54]
  Wk 4 CD8+ effector | -0.90 [-3.58 to 1.38]
  Wk 4 CD8+ immune senescence | -1.83 [-4.05 to 1.10]
  Wk 24 CD8+ total | 2.38 [-1.01 to 4.23]
  Wk 24 CD8+ naive | -0.15 [-2.15 to 0.96]
  Wk 24 CD8+ central memory | 0.75 [-0.45 to 1.78]
  Wk 24 CD8+ effector memory | 0.80 [-0.89 to 2.14]
  Wk 24 CD8+ effector | -2.68 [-7.06 to 1.41]
  Wk 24 CD8+ immune senescence | -3.30 [-8.29 to 0.39]

ADVERSE EVENTS:
Arm/Group | Maraviroc Intensification
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maraviroc Intensification (N=32)
Altered mental status (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-08-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT00925756/Prot_SAP_000.pdf